CLINICAL TRIAL: NCT03822390
Title: Diagnostic Performance of a Convolutional Neural Network for Diminutive Colorectal Polyp Recognition. A Multicentre, Prospective Observational Study
Brief Title: Diagnostic Performance of a Convolutional Neural Network for Diminutive Colorectal Polyp Recognition
Acronym: POLAR
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Bergman Clinics (Other); Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Prof. E. Dekker, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W18_422
Record Dates: First submitted 2019-01-21; First posted 2019-01-30 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Artificial Intelligence; Colorectal Polyp
Keywords: Artificial Intelligence; Computer aided diagnosis; Diminutive colorectal polyps; Optical diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients older than 18 years undergoing colonoscopy in one the participating centres.
  Interventions: Device: CAD-CNN system

INTERVENTIONS:
Device: CAD-CNN system — The CAD-CNN system will be trained in predicting the histology of diminutive polyps. Before training, the dataset will be split up into a training set and a test set. To ensure a completely independent test and training set there will be no overlap between patients (i.e. if polyps from a patient A is present in the training set it cannot be in the test set as well).

SUMMARY:
Rationale: Diminutive colorectal polyps (1-5mm in size) have a high prevalence and very low risk of harbouring cancer. Current practice is to send all these polyps for histopathological assessment by the pathologist. If an endoscopist would be able to correctly predict the histology of these diminutive polyps during colonoscopy, histopathological examination could be omitted and practise could become more time- and cost-effective. Studies have shown that prediction of histology by the endoscopist remains dependent on training and experience and varies greatly between endoscopists, even after systematic training. Computer aided diagnosis (CAD) based on convolutional neural networks (CNN) may facilitate endoscopists in diminutive polyp differentiation. Up to date, studies comparing the diagnostic performance of CAD-CNN to a group of endoscopists performing optical diagnosis during real-time colonoscopy are lacking.

Objective: To develop a CAD-CNN system that is able to differentiate diminutive polyps during colonoscopy with high accuracy and to compare the performance of this system to a group of endoscopist performing optical diagnosis, with the histopathology as the gold standard.

Study design: Multicentre, prospective, observational trial. Study population: Consecutive patients who undergo screening colonoscopy (phase 2)

Main study parameters/endpoints: The accuracy of optical diagnosis of diminutive colorectal polyps (1-5mm) by CAD-CNN system compared with the accuracy of the endoscopists. Histopathology is used as the gold standard.

ELIGIBILITY:
Phase 1A -

- Patients with one polyp subtype (based on histology)

Phase 1B Patients older than 18 years that underwent colonoscopy in one of the participating centres.

Phase 2:- Validation CAD-CNN system

Inclusion Criteria:

All patients older than 18 years old undergoing screenings colonoscopy in one of the participating centres.

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease, Lynch syndrome or (serrated) polyposis syndrome.
* Boston Bowel Preparation Scale (BBPS) <2 in one of the colon segments
* Patients who are unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Phase 1APatients that underwent colonoscopy between 2011-2018 in the Bergman Clinics Amsterdam, in the context of the Dutch bowel cancer screening or surveillance program or because of symptoms.
  Phase 1B Patients older than 18 years that underwent colonoscopy in one of the participating centres.
  Phase 2 All patients older than 18 years old undergoing screenings colonoscopy in one of the participating centres.
Sampling Method: Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
The accuracy of the CAD-CNN system for predicting histology of diminutive colorectal polyps (1-5mm) compared with the accuracy of the prediction of the endoscopist. Both the CAD-CNN system and the endoscopist will use NBI for their predictions. | 2 year
  Accuracy is defined as the percentage of correctly predicted optical diagnoses of the CAD-CNN system and / or endoscopist compared to the gold standard pathology. For the calculation of the accuracy, adenomas and SSLs will be dichotomized as neoplastic polyps, while HPs are considered non-neoplastic

SECONDARY OUTCOMES:
The mean duration in seconds of the CAD-CNN system to make a per polyp diagnosis. | 2 year
  The mean duration in seconds of the CAD-CNN system to make a per polyp diagnosis.
The mean number of attempts of the CAD-CNN to make a diagnosis per polyp | 2 year
  The mean number of attempts of the CAD-CNN to make a diagnosis per polyp
The ratio of unsuccessful diagnosis from all diagnosis of the CAD-CNN system. An unsuccessful diagnosis/failure of the CAD-CNN system is defined as more than 3 unsuccessful attempts | 2 year
  The ratio of unsuccessful diagnosis from all diagnosis of the CAD-CNN system. An unsuccessful diagnosis/failure of the CAD-CNN system is defined as more than 3 unsuccessful attempts
The number of diminutive polyps per colonoscopy that is resected and discarded without histopathological analysis with optical diagnosis strategy (the CAD-CNN system or endoscopist) | 2 year
  The number of diminutive polyps per colonoscopy that is resected and discarded without histopathological analysis with optical diagnosis strategy (the CAD-CNN system or endoscopist)
The percentage of colonoscopies in which diminutive polyps are characterized based on optical diagnosis, removed and discarded without histopathological evaluation (i.e. proportion of polyps assessed with high confidence) | 2 year
  The percentage of colonoscopies in which diminutive polyps are characterized based on optical diagnosis, removed and discarded without histopathological evaluation (i.e. proportion of polyps assessed with high confidence)
The percentage of colonoscopies in which the surveillance interval is based on the optical diagnosis of the CAD-CNN system and the patient can be directly informed of the surveillance interval after colonoscopy | 2 year
  The percentage of colonoscopies in which the surveillance interval is based on the optical diagnosis of the CAD-CNN system and the patient can be directly informed of the surveillance interval after colonoscopy
The percentage of colonoscopies in which diminutive hyperplastic polyps in the rectosigmoid are left in situ. | 2 year
  The percentage of colonoscopies in which diminutive hyperplastic polyps in the rectosigmoid are left in situ.
The diagnostic sensitivity for optical diagnosis of the CAD-CNN system and the endoscopists | 2 year
  The diagnostic sensitivity for optical diagnosis of the CAD-CNN system and the endoscopists
The diagnostic sensitiviy for optical diagnosis of the CAD-CNN system and the endoscopists | 2 year
  The diagnostic sensitiviy for optical diagnosis of the CAD-CNN system and the endoscopists
The accuracy rates on a per polyp basis | 2 year
  Accuracy on a polyp basis is defined as the percentage of correctly predicted optical diagnoses of the CAD-CNN system and / or endoscopist compared to the gold standard pathology. For the calculation of the accuracy on a polyp basis, adenomas, SSLs and HPs are considered different subtypes.
Agreement between recommended surveillance intervals, based on optical diagnosis of diminutive polyps with high confidence, compared to surveillance recommendations based on histology of all polyps | 2 year
  Agreement between recommended surveillance intervals, based on optical diagnosis of diminutive polyps with high confidence, compared to surveillance recommendations based on histology of all polyps
The diagnostic specificity for optical diagnosis of the CAD-CNN system and the endoscopists | 2 year
  The diagnostic specificity for optical diagnosis of the CAD-CNN system and the endoscopists
The diagnostic PPV for optical diagnosis of the CAD-CNN system and the endoscopists | 2 year
  The diagnostic PPV for optical diagnosis of the CAD-CNN system and the endoscopists
The diagnostic NPV for optical diagnosis of the CAD-CNN system and the endoscopists | 2 year
  The diagnostic NPV for optical diagnosis of the CAD-CNN system and the endoscopists

CONTACTS AND LOCATIONS:
Overall Officials: Evelien NA Dekker, Msc, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
There is not yet a plan to share data. However, patients will be asked informed consent with the possibility to share the data.

REFERENCES:
- [Derived] Houwen BBSL, Hazewinkel Y, Giotis I, Vleugels JLA, Mostafavi NS, van Putten P, Fockens P, Dekker E; POLAR Study Group. Computer-aided diagnosis for optical diagnosis of diminutive colorectal polyps including sessile serrated lesions: a real-time comparison with screening endoscopists. Endoscopy. 2023 Aug;55(8):756-765. doi: 10.1055/a-2009-3990. Epub 2023 Jan 9. PMID 36623839
- [Derived] Houwen BBSL, Hartendorp F, Giotis I, Hazewinkel Y, Fockens P, Walstra TR, Dekker E; POLAR study group; *on behalf of the POLAR study group. Computer-aided classification of colorectal segments during colonoscopy: a deep learning approach based on images of a magnetic endoscopic positioning device. Scand J Gastroenterol. 2023 Jun;58(6):649-655. doi: 10.1080/00365521.2022.2151320. Epub 2022 Dec 2. PMID 36458659